CLINICAL TRIAL: NCT03138954
Title: Place of Endoscopic Rectal Ultrasound With Elastosonography and Contrast in Diagnosis and Supported of Deep Pelvic Endometriosis With Bowel Involvement
Brief Title: Endoscopic Rectal UltraSound With Elastosonography and Contrast in Deep Pelvic Endometriosis With Bowel Involvement
Status: Completed | Type: Observational
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, VANBIERVLIET, Head of endoscopy unit, Principal Investigator, Medical Doctorate, Physiology Doctorate, Société Française d'Endoscopie Digestive
Other Study IDs: EEE2018
Record Dates: First submitted 2017-03-30; First posted 2017-05-03 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Endometriosis, Rectum
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study will be to determine the diagnostic and prognostic value of elastosonography and the use of the contrast agent (Sonovue®) in the endoscopic ultrasound exploration of deep pelvic endometriosis.

DETAILED DESCRIPTION:
To diagnose deep infiltrating endometriosis, a clinical examination may be performed by a gynecologist to look for typical signs of endometriosis, but in 25% of case there can be absent.

According to that, medical imaging is indispensable in diagnosis of pelvic endometriosis. Trans vaginal ultrasonography, and pelvic MRI are major tools in the hands of specialists, but several studies have shown the importance of endoscopic rectal ultrasound, with a sensitivity close to 90% for de diagnosis of digestive impairment.

In recent years the use of elastography and the injection of microbubbles of sulfur hexafluoride in addition to endoscopic ultrasound has made it possible to improve the diagnostic accuracy of the technique in tumoral pathologies, in particular bilio-pancreatic injuries.

However, no study has yet evaluated the endoscopic rectal ultrasound with elastometry and injection of contrast agent to characterize the digestive lesions of deep pelvic endometriosis.

The endoscopic rectal ultrasound has demonstrated its place in the evaluation of deep pelvic endometriosis disease but its latest complementary techniques of interest have not yet been studied prospectively. The aim of the study will be to determine the diagnostic and prognostic value of elastosonography and the use of the contrast agent (Sonovue®) in the endoscopic ultrasound exploration of deep pelvic endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Woman over 18 years of age
* Diagnosis of deep pelvic endometriosis (clinical and / or MRI and / or transvaginal ultrasound), defined by penetrating endometriosis lesions in the retroperitoneal space and / or pelvic organ wall at a depth of at least 5 millimeters , with digestive impairment.
* Presenting symptoms of deep pelvic endometriosis disabling and / or fertility difficulties and requiring an exhaustive iconographic assessment.
* Belong to a social security scheme.
* Signature of informed consent.

Exclusion Criteria:

* Without medical contraindication to the realization of a low digestive endoscopy.
* Allergy or hypersensitivity to sulfur hexafluoride or one of the components of Sonovue® (contrast agent used in endoscopy ultrasound).
* Severe heart rhythm disorders.
* Angina unstable.
* Recent Acute Coronary Syndrome.
* Heart Shunt Right - Left.
* Severe pulmonary arterial hypertension (PAH) (defined as PAH > 90 mmHg).
* Acute or severe cardiac insufficiency stage 3 and 4
* Pregnant woman and vulnerable patient population (persons deprived of administrative and / or judicial liberty, and persons under guardianship.
* Mental disability of the subject making participation in the trial impossible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with deep pelvic endometriosis and digestive impairment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Relevance of endoscopic elastosonography for description and characterization of digestive endometriosis lesions, using a ratio of elastonography. | 36 months
  Calculate the average of the endoscopic elastosonography ratios in order to establish the hardness of the endometriosic tissues invading the digestive tract. For each lesion, a ratio of elastosonography will be calculated, averaging three elastometric measurements taken during the examination.
Relevance of EUS contrast for description and characterization of digestive endometriosis lesions. | 36 months
  Determine the contrast agent intake, intensity, start time, and washout time, depending on the location, and the extent of the endometriosis lesion to the digestive tract. Using a scale of intensity of contrast intake (Weak, Moderate, Intense)

SECONDARY OUTCOMES:
Correlation between elastosonography and EUS contrast for clinical criteria using visual analog scale of pain. | 36 months
  The first clinical criteria will be based on each patient's pain, using visual analog scale of pain, from the data collected from each patient by completing a questionnaire during the interview.
Correlation between elastosonography and EUS contrast for clinical criteria using , description of symptoms. | 36 months
  The second clinical criteria will be based on each patient's, type of symptoms. Using the data collected from each patient by completing a questionnaire during the interview.
Correlation between elastosonography and EUS contrast for clinical criteria using scale of analgesic used. | 36 months
  The third clinical criteria will be based on different types of drug therapy used for the pain. Using the data collected from each patient by completing a questionnaire during the interview.
Correlation between elastosonography and EUS contrast for histological criteria. | 36 months
  The histological criteria will be established, after anatomopathological analysis of the operative part, on the hardness of the lesions, and their vascularization.
Surgical criteria | 36 months
  The surgical criteria will be based on the type of surgery, its difficulty, and its possible complications according to Clavien d'Indo's classification.
Establish the safety of use of elastosonography and the endoscopy rectal ultrasound using contrast. | 36 months
  The safety of use of the elastosonography and the endoscopy rectal ultrasound using contrast will be established after statistical analysis of possible side effects attributable to the procedure.Number of participants with medical procedure -related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital L'Archet 2, Nice, France

IPD SHARING:
Plan to Share IPD: No